CLINICAL TRIAL: NCT01690403
Title: An Open-label, Non-randomized, Single Sequence, Two Periods, Four-treatment, Three Parallel Groups Pharmacokinetic Interaction Study of Repeated Oral Doses (Daily or Weekly Regimen) of Rifapentine on ATRIPLA™ (Fixed Dose Combination of Efavirenz, Emtricitabine and Tenofovir Disoproxil Fumarate) Given to HIV+ Patients
Brief Title: Interaction Study to Assess the Pharmacokinetic Interaction of Oral Administration of Rifapentine on ATRIPLA™ in HIV Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: INT12291; U1111-1131-1992 (Other: UTN)
Record Dates: First submitted 2012-09-13; First posted 2012-09-21 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — rifapentine; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- cohort 1 (Experimental): Period 1 (15 days) : ATRIPLA™ Period 2 (21 days) : ATRIPLA™ + oral rifapentine (regimen 1).
  Interventions: Drug: rifapentine (M000473); Drug: EFZ EMT TDF
- cohort 2 (Experimental): Period 1 (15 days) : ATRIPLA™ Period 2 (21 days) : ATRIPLA™ + oral rifapentine (regimen 2).
  Interventions: Drug: rifapentine (M000473); Drug: EFZ EMT TDF
- cohort 3 (optional) (Experimental): Period 1 (15 days) : ATRIPLA™ Period 2 (21 days) : ATRIPLA™ + oral rifapentine (regimen 3).
  Interventions: Drug: rifapentine (M000473); Drug: EFZ EMT TDF

INTERVENTIONS:
Drug: rifapentine (M000473) — Pharmaceutical form:tablet
  Route of administration: oral
Drug: EFZ EMT TDF — Pharmaceutical form:tablet
  Route of administration: oral
  Other Names: ATRIPLA™

SUMMARY:
Primary Objective:

- To evaluate the effect of single and repeated administration of rifapentine given as daily or weekly regimen on steady-state pharmacokinetic parameters of efavirenz, emtricitabine and tenofovir given as a fixed dose combination (ATRIPLA™ ).

Secondary Objective:

- To evaluate the safety and tolerability of concomitant administration of rifapentine and ATRIPLA™ given to HIV+ patients

DETAILED DESCRIPTION:
* Screening to admission: up to 21 days
* Admission to the end of the follow-up: up to 41 days

  * Period 1: Treatment period of 15 days with ATRIPLA™ (background therapy). Patients should receive the same regimen and dose of ATRIPLA™ during the all study screening and period 1.
  * Period 2: Treatment over a period of 21 days in co-administration with rifapentine.
  * Follow up: 3 to 5 days after the last rifapentine administration.

ELIGIBILITY:
Inclusion criteria :

- HIV+ male and female patients receiving ATRIPLA™ aged 18 to 55 years old with a CD4 count cells of at least 350

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, haematological (patients with porphyria), neurological, osteomuscular, articular, psychiatric, systemic, ocular, gynaecologic (if female), or infectious disease, or signs of acute illness other than HIV disease.
* Active or latent tuberculosis infection

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
To determine PK parameters Cmax, Cmin and AUC0-24 for efavirenz (EFZ), emtricitabine (EMT) and tenofovir (TDF) | Day-2, Day 1 and Day 21 for cohorts 1 and 3, and on Day -2 ,Day 1 and Day 16 for cohort 2

SECONDARY OUTCOMES:
To determine PK parameters t1/2z, tmax for efavirenz (EFZ), emtricitabine (EMT) and tenofovir (TDF) | Day-2, Day 1 and Day 21 for cohorts 1 and 3, and on Day -2, Day 1 and Day 16 for cohort 2
To determine PK parameters tlag, CL/F for efavirenz (EFZ), emtricitabine (EMT) and tenofovir (TDF) | Day-2, Day 1 and Day 21 for cohorts 1 and 3, and on Day -2, Day 1 and Day 16 for cohort 2
To determine PK parameter for AUC0-10 for efavirenz (EFZ), emtricitabine (EMT) and tenofovir (TDF) | Day -2 and Day 1 for cohorts 1 and 3
To determine PK parameters Ctrough for rifapentine and 25-desacetyl- rifapentine (25-DR) | Cohort 2: Day 1, 8, and 15
To determine PK parameters C8h for rifapentine and 25-desacetyl- rifapentine (25-DR) | Cohort 2: Day 1, 8, and 15

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 840001, Buffalo, New York, United States